CLINICAL TRIAL: NCT04255355
Title: Comparing the Effects of Pelvic Alignment and Diaphragmatic Breathing on Glenohumeral Internal Rotation Deficit (GIRD) - A Randomized Control Trial
Brief Title: Comparing the Effects of Pelvic Alignment Versus Diaphragmatic Breathing on Shoulder Range of Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of North Georgia (Other)
Responsible Party: Principal Investigator, Mohammad(Reza) Nourbakhsh, Professor, University of North Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 2019-158
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Glenohumeral Internal Rotation Deficit; Pelvic Misalignment; Diaphragmatic Breathing
Keywords: Shoulder; Pelvis; Regional interdependence; Diaphragm

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pelvic alignment and forceful expiration exercise (Active Comparator)
  Interventions: Other: Pelvic alignment and forceful expiration
- Pelvic repositioning exercise (Experimental)
  Interventions: Other: Pelvic repositioning exercise
- Diaphragmatic breathing exercise (Experimental)
  Interventions: Other: Diaphragmatic breathing exercise

INTERVENTIONS:
Other: Pelvic alignment and forceful expiration — The participant will be in supine with feet flat on a wall and the knees and hips flexed to 90 degrees. A standard 5" ball will be placed between the knees. The participant will hold a standard 9-inch balloon in the mouth with one hand. The subject will be instructed to isometrically contract the hamstrings to lift the ischium off the table while maintaining a posterior pelvic tilt. In this position, subject will be instructed to perform isometric hip adduction by squeezing the ball placed between the knees. The subject will then be instructed to breathe in through the nose and blow the air out into the balloon with full exhalation to activate the transverse and oblique abdominals. The participant will hold the breath for 3 seconds while maintaining hamstring contraction, adductor contraction, and transverse and oblique abdominal contraction. This process will be repeated four times. This exercise will be performed once daily under the supervision of the therapist for 5 days.
  Arms: Pelvic alignment and forceful expiration exercise
Other: Pelvic repositioning exercise — The participant will be positioned supine with their feet flat on a wall and the knees and hips flexed to 90 degrees. The subject will be instructed to isometrically contract the hamstrings to allow the ischial tuberosities to lift off the table while also maintaining a posterior pelvic tilt. The tailbone should be slightly lifted off the table, the abdominal muscles should be relaxed, and the low back should be flat on the table. While maintaining the posterior pelvic tilt, the subject will be instructed to perform isometric hip adduction by squeezing the ball that is placed between the knees. The subject will hold for 3 seconds and then relax. This process will be repeated four times. This exercise will be performed daily under the supervision of the therapist for 5 days.
  Arms: Pelvic repositioning exercise
Other: Diaphragmatic breathing exercise — For diaphragmatic breathing exercise, the subject will be in supine position. The investigator places both hands around the participant's lower ribs and abdominal area. The investigator applies slight manual resistance to the chest and abdominal wall during inhalation phase of breathing.The participant is instructed to apply outward pressure against the investigator resistance and to raise the chest and abdominal wall simultaneously with inhalation. Then participants performs a full exhalation and hold his/her breath for 3 seconds before breathing in again. This process is repeated for 4 breathing cycles. Participants will perform this exercise once a day under investigator supervision.
  Arms: Diaphragmatic breathing exercise

SUMMARY:
The goal of this research study is to compare the effects of pelvic alignment versus diaphragmatic breathing on range of motion in the shoulder joint in both athletic and nonathletic population. The investigators plan to have approximately 45 participants to take part in this study. Subjects will be assigned into three groups. Group 1 will perform both pelvic alignment and diaphragmatic breathing exercises. This group will be used as the standard or control group. Group 2 will perform pelvic alignment exercise only; and Group 3 will perform diaphragmatic exercises only. The shoulder internal rotation range will be assessed in all three groups. Maximal expiratory rate will be measured in group 3 to assure improved diaphragmatic breathing in subjects. The shoulder internal rotation range in group 2 & 3 will be compared to the shoulder range of motion in the standard group.

DETAILED DESCRIPTION:
Study design This study is a randomized, blinded, pretest-posttest control group experimental design comparing the effects of pelvic alignment vs. diaphragmatic breathing on Glenohumeral Internal Rotation Deficit (GIRD). Protection of the subjects' rights will be secured through a signed informed consent form approved by the university Institutional Review Board.

Subject selection, randomization, and blinding process: Using statistical power analysis 45 healthy, college aged participants are needed for this study. These subjects will be volunteers and recruited by word of mouth by campus professors, coaches and physical therapy students and faculty.

Intervention timeline: Baseline assessment (pretest), five treatment sessions and a posttest. The time required by subjects will be between five and seven days total with each immediately succeeding the next. Treatment sessions will be approximately 10 minutes each. If any portion of this timeline happens to fall outside of the university operational hours, then the intervention will resume the following day. Subjects will be informed of their rights to receive the results of their assessments following the conclusion of the study. Two of the investigators will perform the initial screenings, groups assignments and treatments for all subjects. The other two investigators, who are blinded on participant's group assignment will perform all pretest and posttest measurements. Intraclass Correlation Coefficient model (3,3) will be used, in a pilot study, to assess inter-rater and intra-rater reliability for all testing procedures.

Testing Procedures:

The primary measurements include Ober's test, assessment of shoulder internal rotation range of motion, and spirometry measurements of maximal expiratory rate.

Range of motion assessment: A Cybex isokinetic table will be used to measure passive shoulder internal rotation range of motion. The Cybex will provide standardized arm position and accurate digital measurement of the shoulder internal rotation bilaterally. All pretest and posttest ROM measurements will be performed by the same examiners.

Pelvic alignment assessment: Ober's test will be used to assess pelvic alignment. Although this test is widely known as an assessment of iliotibial band/fascia lata length, it was originally used to assess pelvic alignment. It has been suggested that a unilateral positive Ober's test is indicative of hemipelvic anterior tilt and forward rotation, which leads to a bony block of the rim of the acetabulum on the femoral neck. This bony block would decrease the amount of adduction, leading to a positive Ober's test.

Craig's test will be used during the screening process to assess presence of excessive femoral anteversion angle.

Spirometry: A digital spirometer is used for measuring maximal expiratory rate.

Treatment Procedures:

Neuromuscular Exercise for combined Pelvic Alignment and Diaphragmatic Breathing:

Pelvic alignment and diaphragmatic breathing exercise included simultaneous activation of the hamstring, hip adductor and transverse abdominal muscles with forceful exhalation.

Pelvic Alignment Exercises: Pelvic alignment involves simultaneous activation of the hamstring muscles and hip adductors to reset pelvic symmetry.

Diaphragmatic Breathing exercise: Diaphragmatic breathing involves subject education for simultaneous rise of chest and abdominal wall with inhalation.

ELIGIBILITY:
Inclusion Criteria

* Having a unilateral positive Ober's test
* Having reduced (more than 15 degrees) shoulder internal rotation in the contralateral shoulder

Exclusion Criteria

* Having a positive Craig's test
* Having bilateral positive Ober's test
* Structural leg length discrepancies
* Having shoulder pain, back pain or any other musculoskeletal pain or dysfunctions
* Having any other medical conditions that prevents them from performing physical exercise
* Having any respiratory or other medical conditions that prevents them from performing deep breathing and expiratory exercises.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-07-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in shoulder internal rotation rang of motion | Change from baseline internal rotation range of motion after 5 days of intervention
  A Cybex isokinetic table will be used for standard positioning of the participants's arm. the participant will be positioned in supine, with his/her arm supported on the dynamometer's arm for shoulder assessment. Shoulder internal rotation range of motion will be assessed using the digital goniometer incorporated into the cybex dynamometer.
Changes in Maximal expiratory rate | Change from baseline expiratory rate after 5 days of intervention
  A digital spirometer (EasyOne Plus Diagnostic Spirometry System) will be use for assessing maximal expiratory rate. A maximal expiratory test will be performed with the subject in sitting. A nose clip will be used to ensure all air is going into the manometer. Our measurements will be taken from total lung capacity, so the subject will first fully inhale, then fully exhale, pausing for 1-2 seconds at the end.

SECONDARY OUTCOMES:
Change in pelvic alignment | Change from baseline hip adduction range of motion after 5 days of interventjion
  Ober's test will be used to assess pelvic alignment. Limited hip joint adduction range of motion is considered as a positive test.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Nourbakhsh, PhD, Principal Investigator — University of North Georgia
Locations (1):
- University of North Georgia, Dahlonega, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the results have been published